CLINICAL TRIAL: NCT03904563
Title: A Single-armed Phase Ⅱ Study of Bevacizumab Maintenance Therapy After Chemoradiotherapy for Locally Advanced Lung Adenocarcinoma
Brief Title: Bevacizumab After Chemoradiotherapy For Locally Advanced Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1046
Record Dates: First submitted 2019-03-13; First posted 2019-04-05 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Lung Adenocarcinoma
Keywords: bevacizumab; Split-course Chemoradiotherapy
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab (Experimental): All patients received four cycles of weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡)(DP), each of 1 day's duration, combined with split-course thoracic radiotherapy, with one-month break.Then every patients are treated with Bevacizumab 1-2 months later.The recommended dose for intravenous infusion is 15mg/kg body weight, which is given every 3 weeks for up to 1 year.
  Interventions: Drug: Bevacizumab; Radiation: chest radiation; Drug: concurrent chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Patients are treated with Bevacizumab 1-2 months after the chemoradiotherapy.The recommended dose for intravenous infusion is 15mg/kg body weight, which is given every 3 weeks for up to 1 year.
Radiation: chest radiation — split-course chest radiation
Drug: concurrent chemotherapy — weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡) concurrent with chest radiation

SUMMARY:
This prospective phase II study is to determine the efficacy and safety of bevacizumab maintenance therapy after concurrent chemoradiotherapy in locally advanced lung adenocarcinoma

DETAILED DESCRIPTION:
This prospective phase II study is to determine the efficacy and safety of bevacizumab maintenance therapy after concurrent chemoradiotherapy in locally advanced lung adenocarcinoma.

All patients received 4 cycles of weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡)(DP), each of 1 day's duration, combined with split-course thoracic radiotherapy, with one-month break.Bevacizumab maintenance therapy starts 1-2 months later after the chemotherapy.The recommended dose for intravenous infusion is 15mg/kg body weight, and the drug is given every 3 weeks for up to 1 year. Toxicities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of lung adenocarcinoma
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Unresectable, refusing surgery or after R2 surgery ,confirmed by PET-CT or chest and abdominal CT, craniocerebral MRI, and ECT.
* After radiotherapy and chemotherapy, the tumor is in partial remission, complete remission or stable.
* 1-2 months after chemoradiotherapy ends.
* Organ and bone marrow functions were normal within the first 30 days of enrollment, including: • AST, ALT≤ 2.5*ULN or ≤5*ULN (with liver metastasis); • TBil ≤ 1.5 ULN • neutrophils absolute value ≥500 cells/mm3 • creatinine clearance ≥45 mL/min ;• platelets≥50,000 cells/mm3.
* CB6 within normal limits
* Patients and their family signed the informed consents

Exclusion Criteria:

* Lung squamous carcinoma.
* The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava).
* The tumor was associated with a cavity over 2cm in diameter.
* Bleeding tendency or coagulation disorder.
* Patients with hemoptysis (1/2 teaspoon blood/day) within 1 month.
* Full-dose anticoagulation therapy was used within the past 1 month.
* Severe vascular disease occurred within 6 months.
* Gastrointestinal fistula, perforation or abdominal abscess occurred within 6 months.
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months.
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg).
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours.
* Urine protein 3-4+, or 24h urine protein quantitative >1g.
* Degree 3 esophagitis after chemoradiotherapy has not recovered.
* Elderly patients (age 75 years).
* The investigator does not consider the participant to be eligible for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3-year
  Progression-free survival in patients
rate of grade≥2 radiation pneumonia(NCI-CTC4.0) | 1 year from the end of chemoradiotherapy
  radiation-induced pulmonary injury is classified into 1-5 grades according to NCI-CTC4.0. The incidence of symptomatic radiation-induced pulmonary injury: the ratio of grade 2 and above radiation-induced pulmonary injury cases in 1 year after radio therapy to all cases can be evaluated .

SECONDARY OUTCOMES:
overall survival | 3-year
  overall survival
response rate | 3-year
rate of grade 3-4 radiation esophagitis | 3-year
rate of grade 3-4 radiation pneumonitis | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Chun SG, Hu C, Choy H, Komaki RU, Timmerman RD, Schild SE, Bogart JA, Dobelbower MC, Bosch W, Galvin JM, Kavadi VS, Narayan S, Iyengar P, Robinson CG, Wynn RB, Raben A, Augspurger ME, MacRae RM, Paulus R, Bradley JD. Impact of Intensity-Modulated Radiation Therapy Technique for Locally Advanced Non-Small-Cell Lung Cancer: A Secondary Analysis of the NRG Oncology RTOG 0617 Randomized Clinical Trial. J Clin Oncol. 2017 Jan;35(1):56-62. doi: 10.1200/JCO.2016.69.1378. Epub 2016 Oct 31. PMID 28034064
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Ahn JS, Ahn YC, Kim JH, Lee CG, Cho EK, Lee KC, Chen M, Kim DW, Kim HK, Min YJ, Kang JH, Choi JH, Kim SW, Zhu G, Wu YL, Kim SR, Lee KH, Song HS, Choi YL, Sun JM, Jung SH, Ahn MJ, Park K. Multinational Randomized Phase III Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-Small-Cell Lung Cancer: KCSG-LU05-04. J Clin Oncol. 2015 Aug 20;33(24):2660-6. doi: 10.1200/JCO.2014.60.0130. Epub 2015 Jul 6. PMID 26150444
- [Background] Tsujino K, Kurata T, Yamamoto S, Kawaguchi T, Kubo A, Isa S, Hasegawa Y, Ou SH, Takada M, Ando M. Is consolidation chemotherapy after concurrent chemo-radiotherapy beneficial for patients with locally advanced non-small-cell lung cancer? A pooled analysis of the literature. J Thorac Oncol. 2013 Sep;8(9):1181-9. doi: 10.1097/JTO.0b013e3182988348. PMID 23883782
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Reck M, von Pawel J, Zatloukal P, Ramlau R, Gorbounova V, Hirsh V, Leighl N, Mezger J, Archer V, Moore N, Manegold C. Phase III trial of cisplatin plus gemcitabine with either placebo or bevacizumab as first-line therapy for nonsquamous non-small-cell lung cancer: AVAil. J Clin Oncol. 2009 Mar 10;27(8):1227-34. doi: 10.1200/JCO.2007.14.5466. Epub 2009 Feb 2. PMID 19188680
- [Background] Zhou C, Wu YL, Chen G, Liu X, Zhu Y, Lu S, Feng J, He J, Han B, Wang J, Jiang G, Hu C, Zhang H, Cheng G, Song X, Lu Y, Pan H, Zheng W, Yin AY. BEYOND: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study of First-Line Carboplatin/Paclitaxel Plus Bevacizumab or Placebo in Chinese Patients With Advanced or Recurrent Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Jul 1;33(19):2197-204. doi: 10.1200/JCO.2014.59.4424. Epub 2015 May 26. PMID 26014294
- [Background] Nadler E, Yu E, Ravelo A, Sing A, Forsyth M, Gruschkus S. Bevacizumab treatment to progression after chemotherapy: outcomes from a U.S. community practice network. Oncologist. 2011;16(4):486-96. doi: 10.1634/theoncologist.2010-0287. Epub 2011 Mar 25. PMID 21441299
- [Background] Gallet P, Phulpin B, Merlin JL, Leroux A, Bravetti P, Mecellem H, Tran N, Dolivet G. Long-term alterations of cytokines and growth factors expression in irradiated tissues and relation with histological severity scoring. PLoS One. 2011;6(12):e29399. doi: 10.1371/journal.pone.0029399. Epub 2011 Dec 22. PMID 22216271
- [Background] Wozniak AJ, Moon J, Thomas CR Jr, Kelly K, Mack PC, Gaspar LE, Raben D, Fitzgerald TJ, Pandya KJ, Gandara DR. A Pilot Trial of Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Docetaxel and the Combination of Bevacizumab (NSC-704865) in Patients With Inoperable Locally Advanced Stage III Non-Small-Cell Lung Cancer: SWOG S0533. Clin Lung Cancer. 2015 Sep;16(5):340-7. doi: 10.1016/j.cllc.2014.12.014. Epub 2015 Jan 9. PMID 25703100
- [Background] Spigel DR, Hainsworth JD, Yardley DA, Raefsky E, Patton J, Peacock N, Farley C, Burris HA 3rd, Greco FA. Tracheoesophageal fistula formation in patients with lung cancer treated with chemoradiation and bevacizumab. J Clin Oncol. 2010 Jan 1;28(1):43-8. doi: 10.1200/JCO.2009.24.7353. Epub 2009 Nov 9. PMID 19901100